CLINICAL TRIAL: NCT01854814
Title: The Effects of Mycophenolate Mofetil on Renal Outcomes in Patients With Advanced IgA Nephropathy: a Randomized Open-label Study
Brief Title: The Effects of Mycophenolate Mofetil (MMF) on Renal Outcomes in Advanced Immunoglobulin A (IgA) Nephropathy Patients
Acronym: MAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fan Fan Hou (Other)
Responsible Party: Sponsor-Investigator, Fan Fan Hou, Chief of Division of Nephrology, Nanfang Hospital, Southern Medical University
Organization: Nanfang Hospital, Southern Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAIN
Record Dates: First submitted 2013-05-09; First posted 2013-05-16 (Estimated); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Mycophenolic Acid; Losartan

ARMS (2):
- mycophenolate mofetil (Experimental): mycophenolate mofetil 1.5g/day and maximum tolerated labeled dose of losartan
  Interventions: Drug: Mycophenolate mofetil
- losartan (Active Comparator): maximus tolerated labeled dose of losartan
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Mycophenolate mofetil — Mycophenolate mofetil 1.5g/day plus maximum tolerated labeled dose losartan
  Arms: mycophenolate mofetil
Drug: Losartan — Maximum tolerated labeled dose of Losartan
  Arms: losartan

SUMMARY:
The study is to evaluate the effect of Mycophenolate Mofetil compared with losartan alone on time to doubling of serum creatinine or the onset of end stage renal disease in patients with advanced IgA nephropathy who are treated with the maximal tolerated daily dose of losartan.The study will also assess the effects of MMF compared with losartan alone on the changes of urine albumin excretion and the changes in estimated glomerular filtration rate.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven primary IgA nephropathy with urinary proteinuria excretion over 1g/24 hour,subjects must meet 2 of the following criteria:

  1. global glomerular sclerosis plus focal segmental glomerular sclerosis ratio ≥50%
  2. eGFR 30 to 60 ml/min
  3. Hypertension (blood pressure over 140/90 mmHg or taking antihypertensive drugs)

Exclusion Criteria:

1. Secondary IgA nephropathy
2. Familial IgA nephropathy
3. Concomitant disease: cancer, infection, diabetes mellitus, connective tissue disease, abnormal liver function
4. Pregnancy or breasting
5. Inability to comply with study and follow-up procedures

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2022-02 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of mycophenolate mofetil on a composite renal outcomes in subjects with advanced IgA nephropathy | 3 years
  Time to the first occurrence of a component of the composite renal endpoint:
  Doubling of serum creatinine or the onset of end stage renal disease (ESRD) [needing chronic dialysis or renal transplantation or renal death]
To evaluate the effects of mycophenolate mofetil on progression of CKD in subjects with advanced IgA nephropathy | 3 years
  A decrease in eGFR of 30% or more and to a level of less than 60 ml/min at the exit visit if the baseline eGFR was 60 ml/min or more.
  Or a decrease in eGFR of 50% or more at the exit visit if the baseline eGFR was less than 60 ml/min.

SECONDARY OUTCOMES:
To evaluate the effects of mycophenolate mofetil on the changes of proteinuria in subjects with advanced IgA nephropathy | 3 years
  Changes of urinary protein excretion rate
To evaluate the effects of mycophenolate mofetil rapid progression of CKD in subjects with advanced IgA nephropathy | 3 years
  Time to 30% reduction in estimated glomerular filtration rate (eGFR); eGFR reduction greater than 5 ml/min/1.73m^2/year

CONTACTS AND LOCATIONS:
Overall Officials: Fan Fan Hou, M.D., PhD, Principal Investigator — Division of nephrology, Nanfang Hospital Southern Medical University
Locations (3):
- China (3):
  - Nanfang Hospital Southern Medical University, Guangzhou, Guangdong
  - The Fourth People's Hospital Shenzhen, Shenzhen, Guangdong
  - The Institute of Nephrology, Guangdong Medical College, Zhanjiang, Guangdong

REFERENCES:
- [Background] Tang SC, Tang AW, Wong SS, Leung JC, Ho YW, Lai KN. Long-term study of mycophenolate mofetil treatment in IgA nephropathy. Kidney Int. 2010 Mar;77(6):543-9. doi: 10.1038/ki.2009.499. Epub 2009 Dec 23. PMID 20032964
- [Background] Frisch G, Lin J, Rosenstock J, Markowitz G, D'Agati V, Radhakrishnan J, Preddie D, Crew J, Valeri A, Appel G. Mycophenolate mofetil (MMF) vs placebo in patients with moderately advanced IgA nephropathy: a double-blind randomized controlled trial. Nephrol Dial Transplant. 2005 Oct;20(10):2139-45. doi: 10.1093/ndt/gfh974. Epub 2005 Jul 19. PMID 16030050
- [Derived] Alladin A, Hahn D, Hodson EM, Ravani P, Pfister K, Quinn RR, Samuel SM. Immunosuppressive therapy for IgA nephropathy in children. Cochrane Database Syst Rev. 2024 Jun 12;6(6):CD015060. doi: 10.1002/14651858.CD015060.pub2. PMID 38864363
- [Derived] Hou FF, Xie D, Wang J, Xu X, Yang X, Ai J, Nie S, Liang M, Wang G, Jia N; MAIN Trial Investigators. Effectiveness of Mycophenolate Mofetil Among Patients With Progressive IgA Nephropathy: A Randomized Clinical Trial. JAMA Netw Open. 2023 Feb 1;6(2):e2254054. doi: 10.1001/jamanetworkopen.2022.54054. PMID 36745456